CLINICAL TRIAL: NCT01660958
Title: Innovative Strategies to Promote Early Child Development Among Low-income Rural Infants and Preschoolers in India Through Multiple Micronutrient Fortification and Early Learning Opportunities
Brief Title: Project Grow Smart: Intervention Trial of Multiple Micronutrients and Early Learning Among Infants in India
Acronym: GrowSmart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Indian Council of Medical Research (Other Government); The Mathile Institute for the Advancement of Human Nutrition (Other); Micronutrient Initiative (Other)
Responsible Party: Principal Investigator, Maureen Black, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 00048720
Record Dates: First submitted 2012-07-26; First posted 2012-08-09 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Nutritional Deficiencies; Developmental Delay
Keywords: Micronutrient Deficiencies; Early Child Development; Infant Growth; Iron Deficiency
MeSH Terms: conditions — Malnutrition; Learning Disabilities; Iron Deficiencies | interventions — Growth and Development

STUDY DESIGN:
Intervention Model Description: * The infant phase is a factorial design.
  * The preschool phase is a cluster-randomized trial (MNP/placebo nested within high/low-quality preschools).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Infants: MNP (Experimental): • Infants will receive sachets of multiple micronutrient powder (MNP) vs. placebo.
  Interventions: Dietary Supplement: MNP
- Infants: Early Learning (Experimental): • Infant will receive early learning messages delivered in the home by village level workers vs. routine care.
  Interventions: Behavioral: Early Learning
- Infants: No intervention (No Intervention): * Placebo intervention include exposure to a single vitamin (B2 or riboflavin), plus the filler (maltodextrin).
  * Infant phase. Routine care - no early learning intervention
- Infants: MNP/Early Learning (Experimental): * Infants receive the MNP plus early learning intervention by receiving MNP sachets
  * Caregivers receive early learning messaged delivered at home biweekly for one year
  Interventions: Dietary Supplement: MNP; Behavioral: Early Learning
- Preschoolers:MNP/High qual preschool (Experimental): * Preschoolers will receive MNP fortified food in their Anganwadi Centers at the mid-day meal.
  * Preschool quality will be assessed through observations using the Indian-modified ECERS and HOME Inventory for preschools. Using a median split, preschools will be classified as high/low quality. Using a randomization procedure, MNP vs. placebo will be assigned, nested within high/low-quality preschools.
  * Preschools that are classified as high quality preschools.
  Interventions: Dietary Supplement: MNP
- Preschoolers:Placebo/High qual preschool (No Intervention): * Placebo intervention include exposure to a single vitamin (B2 or riboflavin), plus the filler (maltodextrin).
  * Preschool quality will be assessed through observations using the Indian-modified ECERS and HOME Inventory for preschools. Using a median split, preschools will be classified as high/low quality. Using a randomization procedure, MNP vs. placebo will be assigned, nested within high/low-quality preschools.
  * Preschools that are classified as high quality preschools.
- Preschoolers:MNP/Low qual preschool (Experimental): * Preschoolers will receive MNP fortified food in their Anganwadi Centers at the mid-day meal.
  * Preschool quality will be assessed through observations using the Indian-modified ECERS and HOME Inventory for preschools. Using a median split, preschools will be classified as high/low quality. Using a randomization procedure, MNP vs. placebo will be assigned, nested within high/low-quality preschools.
  * Preschools that are classified as low quality preschools.
  Interventions: Dietary Supplement: MNP
- Preschoolers:Placebo/Low qual preschool (No Intervention): * Placebo intervention include exposure to a single vitamin (B2 or riboflavin), plus the filler (maltodextrin).
  * Preschool quality will be assessed through observations using the Indian-modified ECERS and HOME Inventory for preschools. Using a median split, preschools will be classified as high/low quality. Using a randomization procedure, MNP vs. placebo will be assigned, nested within high/low-quality preschools.
  * Preschools that are classified as low quality preschools.

INTERVENTIONS:
Dietary Supplement: MNP — The formulation of the multiple micronutrient powder (MNP) was based on low micronutrient intake, low bioavailability of iron and zinc in the Indian diet, and current World Health Organization (WHO)and Indian recommendations regarding fortification and age-specific nutrient requirements. The MNP formulations were produced by a certified company in India and include: Iron, Vitamin A, Vitamin C, Folic Acid, Zinc, Vitamin B12 Vitamin B2, plus filler (maltodextrin). Placebo included riboflavin and maltodextrin.
  Arms: Infants: MNP; Infants: MNP/Early Learning; Preschoolers:MNP/High qual preschool; Preschoolers:MNP/Low qual preschool
Behavioral: Early Learning — • Infant will benefit from interventions that are based on responsive parenting, whereby caregivers respond to children's cues, provide opportunities for exploration, and engage in nurturant and reciprocal communication.
  Other Names: Care for Development
  Arms: Infants: Early Learning; Infants: MNP/Early Learning

SUMMARY:
Project Grow Smart evaluates the impact fortification with multiple micronutrient powders (MNP) vs. placebo (one vitamin) on child development (primary outcome) and on micronutrient status, growth, and morbidity (secondary outcomes) among young children in rural India (Nalgonda district of Telegana). There is an infant phase and a preschool phase; investigators, study team members, and participants are unaware of whether the fortification is MNP vs. placebo.

The infant phase (enrollment age: 6-14 months) is a 4-cell factorial randomized trial (MNP vs. placebo and early learning vs. routine care), conducted through home visits. Sachets (MNP/placebo) are distributed to be mixed with food. The hypotheses in the infant phase are: 1) MNP leads to better development, growth, and micronutrient status; 2) Early learning leads to better development; 3) Integrated MNP plus early learning leads to better development through both additive and synergistic processes. Developmental evaluations and anthropometric measurements are conducted at baseline, mid-line (6 months), and end-line (12 months). Blood draws for micronutrient status are performed at baseline and endline. Morbidity measures are collected monthly using a morbidity form, modeled after the Demographic and Health Survey.

The preschool phase (enrollment age: 30-48 months) is conducted in Anganwadi Centers (AWC) (preschools). AWC are classified as high or low stimulation, based on an objective observational rating system of the physical environment of the preschools and teacher-child interactions. Preschools are categorized into high/low-quality based on median split, followed by random assignment of MNP/placebo nested within high/low-quality preschools. The hypotheses in the preschool phase are: 1)MNP leads to better development, growth, and micronutrient status; 2) the effect of the MNP on preschoolers' development varies by the quality of the AWC, with stronger effects among preschoolers in high-quality AWCs. The intervention has been modified to coincide with the academic term (September-May). Evaluations are conducted at baseline (September) and end-line (prior to May), with an 8-month intervention period.

DETAILED DESCRIPTION:
Project Grow Smart has two phases: an infant phase and a preschool phase. The design of the two phases differs, although both evaluate the impact of fortification with multiple micronutrient powders (MNP) vs. placebo on child development.

In the infant phase, 6-14 month old infants are recruited and randomized into one of four cells to receive: placebo, placebo plus early learning, MNP alone, and MNP plus early learning (integrated intervention). Interventions are delivered through biweekly (twice/month) home visits by Village Level Workers. Families of all infants receive information on iron rich foods.

The preschool phase is conducted in 22 Anganwadi Centers (AWC) (i.e., preschools). AWC quality is assessed, based on a 109-item observation scale, organized into 18 categories, based on two validated scales: Early Childhood Environment Rating Scale-Revised (ECERS-R) and HOME Inventory, modified to rate the quality of learning opportunities and teacher-child interactions. After training and establishing inter-rater reliability, two psychologists spend four hours in each preschool and independently complete the observation. Scores are summed and averaged. Based on a median split, preschools are categorized into high/low-quality with random assignment of MNP/placebo nested within high/low-quality preschools. Classifications are unknown by investigators, study team, or preschools.

The preschool protocol has been modified to ensure that the trial coincides with the academic term (September-May) to avoid losing the oldest children who transfer to private or primary schools. Baseline evaluations are conducted in September and end-line evaluations are conducted prior to May. Mid-line evaluations have been eliminated. The intervention is delivered over 8 months. The MNP/placebo was supplied to preschools in identical packets of 200 grams, including two measuring spoons of 1 and 0.5 grams. Each packet includes a manufacturer-assigned alphabetic code. AWC workers mix the MNP/placebo into the first bites of the preschoolers' mid-day meal. Mothers receive information on iron-rich food.

ELIGIBILITY:
Inclusion Criteria:

* Participating children must be in one of two age groups: infants: 6-14 months or preschoolers: 30-48 months, inclusive, at time of recruitment.
* Participants must reside in the Nalgonda district of Telengana, India.
* Preschoolers must attend an Anganwadi Center (preschool) in the Nalgonda district that is participating in Project Grow Smart.
* Participating caregivers must be at least 18 years of age at the time of recruitment.

Exclusion Criteria:

* Children with chronic diseases, developmental disabilities, mental retardation, or severe physical handicaps will be excluded
* Children with severe stunting ( <= -3 standard deviation of length-for-age z-score) or severe anemia (hemoglobin < 7 g/dl) will be excluded and referred to a local hospital for evaluation and intervention, as needed..

Ages: 6 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 834 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Infants: Change in cognitive, language, motor, and socio-emotional development | Baseline, Mid-Point (6mo post BL), and End-Point (12mo post BL)
  Data on infants' cognitive, language, motor, and socio-emotional development will be collected at baseline, the 6 month follow-up evaluation, and the 12-month follow-up evaluation using the Mullens Scales of Early Learning.
Preschoolers: Change in cognitive, language, motor, and socio-emotional development | Baseline and End-Point (8mo post BL)
  Data on preschoolers' cognitive, language, motor, and socio-emotional development will be collected at baseline and the 8-month follow-up evaluation using the Mullens Scales of Early Learning.

SECONDARY OUTCOMES:
Infants: Change in micronutrient Status | Baseline and End-Point (12 mo post-baseline)
  Data on infants' micronutrient status (serum ferritin, transferrin receptor, serum zinc, C-reactive protein) and hemoglobin will be collected at baseline and the 12-month follow-up evaluation.
Preschoolers: Change in micronutrient Status | Baseline and End-Point (8mo post BL)
  Data on preschoolers' micronutrient status (serum ferritin, transferrin receptor, serum zinc, C-reactive protein) and hemoglobin will be collected at baseline and the 8-month follow-up evaluation.
Infants: Change in weight and height | Baseline, Mid-Point (6mo post BL), and End-Point (12mo post BL)
  Data on infants' weight and height will be collected at baseline, the 6 month follow-up evaluation, and the 12-month follow-up evaluation
Preschoolers: Change in weight and height | Baseline and End-Point (8mo post BL)
  Data on preschoolers' weight and height will be collected at baseline and the 8-month follow-up evaluation
Infants: Morbidity | Baseline and once a month (for 12mo post BL)
  Morbidity measures (acute respiratory infection and diarrhea) are conducted monthly using a morbidity form, modeled after the Demographic and Health Survey.
Preschoolers: Morbidity | Baseline and once a month (for 8mo post BL)
  Morbidity measures (acute respiratory infection and diarrhea) are conducted monthly using a morbidity form, modeled after the Demographic and Health Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen M Black, PhD, Principal Investigator — University of Maryland, Baltimore; Madhavan K. Nair, PhD, Principal Investigator — NATIONAL INSTITUTE OF NUTRITION
Locations (1):
- National Institute of Nutrition, Hyderabad, Andhra Pradesh, India

REFERENCES:
- [Derived] Black MM, Fernandez-Rao S, Nair KM, Balakrishna N, Tilton N, Radhakrishna KV, Ravinder P, Harding KB, Reinhart G, Yimgang DP, Hurley KM. A Randomized Multiple Micronutrient Powder Point-of-Use Fortification Trial Implemented in Indian Preschools Increases Expressive Language and Reduces Anemia and Iron Deficiency. J Nutr. 2021 Jul 1;151(7):2029-2042. doi: 10.1093/jn/nxab066. PMID 33880548